CLINICAL TRIAL: NCT00002280
Title: An Open Label Study Regimen of Videx (2',3'-Dideoxyinosine, ddI) in Children With Acquired Immunodeficiency Syndrome (AIDS) Who Have Demonstrated Significant Deterioration or Intolerance to Zidovudine (Retrovir)
Brief Title: A Study of ddI in Children With AIDS Who Have Not Had Success With Zidovudine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Masking: None | Purpose: Treatment
Other Study IDs: 039C; AI454-904
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections
Keywords: Didanosine; Drugs, Investigational; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
The purpose of this study is to make didanosine (ddI) available to children with AIDS who are clinically deteriorating on zidovudine (AZT) or intolerant to AZT and cannot enter the Phase II ddI programs due to protocol exclusion or geographic location.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Concomitant medications for the treatment of complications of AIDS.
* CAUTION:
* Concomitant use of ddI with the following drugs must be done with extreme caution:
* Other nucleosides (e.g., ganciclovir).
* Drugs with toxicities similar to those observed with ddI (e.g., phenytoin).
* Drugs with significant pancreatic toxicities, including many drugs used for treatment of major opportunistic infections.
* Use of Sulfonamides or intravenous pentamidine for treatment of acute Pneumocystis carinii pneumonia (PCP) requires discontinuation of ddI for a week following treatment of PCP.
* Caution should also be exercised with patients having intractable diarrhea or patients following a low sodium diet.

Patients must have the following:

- Diagnosis of AIDS. Demonstrated either significant deterioration despite parenteral dosing with zidovudine (AZT) or significant intolerance to AZT.

Signed informed consent by parent or legal guardian. Evaluations every 7-14 days while taking ddI for the first 4 months. Monthly follow-up is required thereafter.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Acute pancreatitis or any history of pancreatitis.
* Seizures or a history of seizure disorder.
* Grade I or greater peripheral neuropathy.
* Preexisting cardiomyopathy.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Chemotherapy with cytotoxic agents.
* AVOID:
* Those agents that may cause pancreatitis such as:
* Pentamidine.
* Sulfonamides.
* Antituberculosis drugs.
* Cimetidine.
* Ranitidine.
* Corticosteroids.
* NOTE the cautionary statement in Patient Inclusion Concurrent Medication.

Patients with the following are excluded:

* Acute pancreatitis or any history of pancreatitis.
* Seizures or a history of seizure disorder.
* Grade I or greater peripheral neuropathy.
* Preexisting cardiomyopathy.

Prior Medication:

Excluded within 15 days of study entry:

* Any anti-retroviral except zidovudine (AZT).

Required:

* Zidovudine (AZT).

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 1994-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol - Myers Squibb Co, Wallingford, Connecticut, United States